CLINICAL TRIAL: NCT03101553
Title: Computerized Treatment for Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016.20077
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpretation Bias Modification (Experimental): Treatment consists of eight brief sessions consisting of two tasks. In Task 1, participants read unique scenarios ("You notice someone pointing in your direction"). A sentence meant to resolve the ambiguity will appear ("This person thinks they reco_nize you"). After filling in the missing letter, the interpretation is reinforced by requiring the participants to correctly answer "yes" or "no" to a comprehension question ("Is this person mocking you?"). In Task 2, participants are shown a word denoting a threatening ("mocking") or benign ("cheerful") interpretation. Participants are presented with an ambiguous scenario ("You hear people at a nearby table laughing") and asked to denote whether the word and the sentence are related. Participants will receive feedback based on their response.
  Interventions: Behavioral: Interpretation Bias Modification
- Progressive Muscle Relaxation (Active Comparator): Participants will receive eight brief sessions of PMR. They will listen to a PMR script (Kassinove & Tafrate, 2002). Participants will be asked to make sure they are sitting comfortably, close their eyes, and systematically tense and release different muscle groups.
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Interpretation Bias Modification — Eight 10-25 minute sessions of interpretation modification to reduce negative interpretation biases related to negative evaluation.
  Arms: Interpretation Bias Modification
Behavioral: Progressive Muscle Relaxation — Eight 15-minute sessions of progressive muscle relaxation (PMR).
  Arms: Progressive Muscle Relaxation

SUMMARY:
The present study aims to examine the feasibility of a computerized treatment for social anxiety disorder. To evaluate the efficacy of the IBM protocol the investigators have developed in reducing evaluation and social threat biases, they will conduct a two-arm randomized controlled trial. Individuals with a diagnosis of social anxiety disorder (N = 50) will be randomized to one of two conditions: 1) IBM or 2) progressive muscle relaxation. Each condition will consist of eight 25 minute treatment sessions. Participants will complete two sessions per week for four weeks and will be administered assessments at pre-treatment, one week post-treatment and at 3-month follow-up. It is hypothesized that: 1) IBM will lead to greater reductions in social anxiety symptoms than the PMR condition; 2) IBM will lead to greater reductions in depression and anxiety than the PMR condition; 3) IBM will lead to greater reductions in threat interpretations and greater increases in benign interpretations than the PMR condition; 4) The effects of condition on social anxiety symptoms will be mediated by changes in social anxiety-related interpretation bias; and 5) The effects of condition will be maintained at the 3-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Social Anxiety Disorder according to DSM-5 criteria
* SPIN score greater than or equal to 30
* Must report sufficient motivation to complete treatment (i.e., score of at least 5 on a 10 point scale (0 = no motivation and 10 = extreme motivation))

Exclusion Criteria:

* Concurrent psychotherapy or treatment for social anxiety disorder
* Clinically significant suicidality
* Current Alcohol Use Disorder of "Severe" severity or higher
* Current Non-alcohol Substance Use Disorder of "Moderate" severity or higher
* Recent changes (less than four weeks) in psychiatric medication
* History of psychotic symptoms
* May not have participated in a similar computerized treatment program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Social Phobia Inventory (SPIN; Davidson, 1995) | change from baseline at one-week post treatment and 3-months post-treatment
  Measures past-week social anxiety symptom severity

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II; Beck, Steer, & Brown, 1996) | change from baseline at one-week post treatment and 3-months post-treatment
  Measures depressive symptom severity
Beck Anxiety Inventory (BAI; Steer & Beck, 1997) | change from baseline at one-week post treatment and 3-months post-treatment
  Measure anxious symptom severity
Interpretations Questionnaire-modified (IQ-modified; Buhlmann et al., 2002) | change from baseline at one-week post treatment and 3-months post-treatment
  Measure of strength of evaluation related threat interpretation bias

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States